CLINICAL TRIAL: NCT04161573
Title: A Preliminary Study on Irony Comprehension Ability of Chinese Speaking Patients With Traumatic Brain Injury
Brief Title: Irony Comprehension Ability of Chinese Speaking Patients With TBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201908029RINA
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Traumatic Brain Injury
Keywords: Irony comprehension
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- TBI group: 15 people in this group. Each should be post TBI for 6 months.
  Interventions: Behavioral: Watching ironic stories
- Control group to TBI: 15 people in this group. Their gender and age accord with TBI group.
  Interventions: Behavioral: Watching ironic stories
- Aging group 1- 20 to 39: Normal people whose age range from 20 to 39.
  Interventions: Behavioral: Watching ironic stories
- Aging group 2- 40 to 59: Normal people whose age range from 40 to 59.
  Interventions: Behavioral: Watching ironic stories
- Aging group 3- above 60: Normal people whose age are above 60.
  Interventions: Behavioral: Watching ironic stories

INTERVENTIONS:
Behavioral: Watching ironic stories — All the participants would be asked to watch a series of self-made stories which are figurative or literal. They have to figure out what is the real meaning of the character's statement. The whole procedure will be done with a computer.

SUMMARY:
This study aims at understanding irony comprehension ability of Chinese speaking patients with TBI through a series of self-made stories. Each story contains two characters having a conversation, and one of them would give a figurative (which is, ironic) or literal statement at the end of the story. The participants are asked to figure out its meaning.

DETAILED DESCRIPTION:
The investigator plans to recruit TBI patients and control group whose gender and age accord with them, 15 people in each group. They would be asked to read the materials mentioned above displaying by a computer. It may take 30 minutes per time, and every participants only do once.

ELIGIBILITY:
Inclusion Criteria:

* Above 20 years old
* Chinese speaking people
* Diagnosed as TBI patients for over 6 months
* Having no other neurological and mental related problems
* Able to read with or without assistive device like glasses

Exclusion Criteria:

* Addicted to alcohol or drug morbid and postmorbid
* Having any communication disorders

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NTUH
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
TBI group gets lower scores | 2 months
  We assume that TBI group can't comprehend ironic statement as well as their control group. Therefore, they may get lower score than their normal- health control group.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chun Chih, PhD, Study Chair — Chung Shan Medical University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Angeleri R, Bosco FM, Zettin M, Sacco K, Colle L, Bara BG. Communicative impairment in traumatic brain injury: a complete pragmatic assessment. Brain Lang. 2008 Dec;107(3):229-45. doi: 10.1016/j.bandl.2008.01.002. Epub 2008 Feb 11. PMID 18267340
- [Result] Carlomagno S, Giannotti S, Vorano L, Marini A. Discourse information content in non-aphasic adults with brain injury: a pilot study. Brain Inj. 2011;25(10):1010-8. doi: 10.3109/02699052.2011.605097. PMID 21812587